CLINICAL TRIAL: NCT06099041
Title: ND-YAG Laser Iris Depigmentation for Cosmoses
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We found complications, intra ocular pressure elevation and iridocyclitis endangered the patients vision
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Elshimaa A.Mateen, Clinical professor, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NILES-EC-CU 23/7/15
Record Dates: First submitted 2023-09-06; First posted 2023-10-25 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Iris Depigmentation
Keywords: Nd-YAG Laser; Iris; Cosmoses
MeSH Terms: interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ND-YAG Laser for iris depigmentation (Other): ND-YAG Laser for iris depigmentation
  Interventions: Device: Nd-YAG Laser for iris depigmentation

INTERVENTIONS:
Device: Nd-YAG Laser for iris depigmentation — Nd-YAG Laser for iris depigmentation

SUMMARY:
Nd-YAG Laser for changing iris coloration by the principle of depigmentation for cosmoses Is that procedure safe or not a prospective study

DETAILED DESCRIPTION:
Nd-YAG Laser for changing iris coloration by the principle of depigmentation for cosmoses Is that procedure safe or not a prospective study safety will be assessed by measuring IOP using Goldman applanation tonometry pre and post-session.

visual acuity assessment in Log-Mar pre and post-session. Refraction assessment pre and post-session. Lens and fundus assessments on slit-lamp and using auxiliary lens 78D

ELIGIBILITY:
Inclusion Criteria:

* clear cornea
* clear lens
* normal IOP < 20 mmHg
* adults aged more than 18 years old
* normal fundus
* dark pigmented iris (black or brown)

Exclusion Criteria:

* Glaucomatous patients and those receiving anti-glaucoma treatment.
* corneal or lens opacity.
* any fundus abnormality

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Monitoring intra-ocular pressure (IOP) by the standard Goldman applanation tonometer before and after ND-YAG Laser for iris depigmentation | one year
  Session of Nd-YAG Laser targeting the iris using power less than that used for peripheral iridotomy causing pigment bleaching to change the iris colour for cosmoses, which may cause pigmentary glaucoma (secondary open angle glaucoma).
Safety of ND-YAG Laser, by visual acuity assessment in log-mar subjectively by using Snellen chart before and after ND-YAG Laser | one year
  If ND-YAG LASER could affect visual acuity.

CONTACTS AND LOCATIONS:
Locations (1):
- Elshimaa A.Mateen, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided